CLINICAL TRIAL: NCT07299656
Title: Outcome of Active Aspiration Versus Simple Compression to Remove Residual Gas From Abdominal Cavity in Reducing Pain After Laparoscopic Cholecystectomy
Acronym: Lap Chole
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: King Edward Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Kemu/draizaztariq
Record Dates: First submitted 2025-12-10; First posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Shoulder Pain; Abdominal Pain (AP)
Keywords: abdominal pain; shoulder pain; laparoscopic procedure; cholecystectomy; pneumoperitonium; lap chole; laparoscopic cholecystectomy
MeSH Terms: conditions — Shoulder Pain; Abdominal Pain

STUDY DESIGN:
Intervention Model Description: Study Design: Comparative study Setting: East Surgical Ward, Mayo Hospital, Lahore. Duration of Study: Six months after approval of synopsis. Sample Size: 62 cases in each group were calculated by taking 5 % level of significance and 80% power of study with expected population proportion of analgesics requirement 43.2% in active gas aspiration group versus 67.6% in simple compression group (p value < 0.001). [9] Sampling Technique: Simple random sampling technique
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group B (Simple compression) (Placebo Comparator): In this group, diagnostic laparoscopies commenced with a 5 mm intraumbilical vertical incision, followed by placement of the first bladeless umbilical port trocar (using 5 mm XCEL). Warm CO2 gas insufflation will create the pneumoperitoneum at a flow rate of 1-2.5 L/min; intra-abdominal pressure will be set at 12 mmHg. Patients will then placed in the Trendelenburg position (45°) and the second trocars (using 5 mm XCEL) will be placed at the suprapubic area. Chromopertubation with methylene blue will be performed, with electrocauterization of the endometriotic lesions if necessary. CO2 insufflation will be then ceased and all trocars will be opened. The surgeon will apply abdominal pressure to evacuate any residual CO2. The patient will be then placed in a neutral (horizon plane) position, the trocars will be removed and the incision closed.
  Interventions: Behavioral: simple compression
- Group A (Active gas aspiration) (Active Comparator): Active Gas Aspiration: Once the trocars will be opened, aspiration cannula will be then placed through the accessory port reach at the subdiaphragmatic under direct visualization. After cessation of CO2 insufflation, residual gas will be removed by suctioning with 100 mmHg of pressure until the infra-diaphragmatic area of the abdominal wall close to liver surface. Negative pressure will be then ceased and the aspiration cannula will be taken out under direct vision. The procedure will be completed using the same method as the simple compression group.
  Interventions: Procedure: Group A (Active Aspiration)

INTERVENTIONS:
Procedure: Group A (Active Aspiration) — Once the trocars will be opened, aspiration cannula will be then placed through the accessory port reach at the subdiaphragmatic under direct visualization. After cessation of CO2 insufflation, residual gas will be removed by suctioning with 100 mmHg of pressure until the infra-diaphragmatic area of the abdominal wall close to liver surface. Negative pressure will be then ceased and the aspiration cannula will be taken out under direct vision. The procedure will be completed using the same method as the simple compression group.
  Arms: Group A (Active gas aspiration)
Behavioral: simple compression — Active Gas Aspiration: Once the trocars will be opened, aspiration cannula will be then placed through the accessory port reach at the subdiaphragmatic under direct visualization. After cessation of CO2 insufflation, residual gas will be removed by suctioning with 100 mmHg of pressure until the infra-diaphragmatic area of the abdominal wall close to liver surface. Negative pressure will be then ceased and the aspiration cannula will be taken out under direct vision. The procedure will be completed using the same method as the simple compression group.
  Arms: Group B (Simple compression)

SUMMARY:
The aim of this study is to compare outcome of active aspiration versus simple compression to remove residual gas from abdominal cavity in reducing pain after laparoscopic cholecystectomy.

DETAILED DESCRIPTION:
INTRODUCTION: Laparoscopic cholecystectomy (LC) is superior to open cholecystectomy for a number of reasons: it causes less discomfort to the patient, reduces the length of the hospital stay, minimizes wound problems, promotes the speedy postoperative return to former activities and causes fewer postoperative pulmonary complications.[1,2] However, disturbing abdominal and shoulder pain can be observed after laparoscopic surgery. The elimination or reduction of this pain may increase patient comfort, promote a quick return to normal activity and reduce pulmonary and venous system problems.[3,4] In studies performed in the 1980s, Riedel and Semm showed radiologically that carbon dioxide (CO2 ) gas remained in the peritoneal area following abdominal laparoscopy.[5] Several studies indicate that this gas leads to irritation and shoulder pain if it remains below the diaphragm following laparoscopy.[6] However, pain after laparoscopy is multifactorial and can be associated with many issues: abdominal muscle tension in the abdominal front wall caused by pneumoperitoneum (Pp); the temperature and volume of insufflated gas; anaesthetic drugs and their postoperative effects; wound size; and the use of intraperitoneal acid during the operation.[7-8] A study aimed to evaluate the effectiveness of active gas aspiration to reduce postoperative shoulder pain in patients undergoing laparoscopy. The shoulder pain scores of the active gas aspiration group showed lower pain intensity than the simple gas evacuation group, with statistically significant results at all time points. There was no significant difference in surgical wound pain. The proportion of patients who required postoperative rescue analgesics was lower in the study than in control group (43.2% vs 67.6%, P = 0.035). There was no significant difference in adverse events until 24 h after surgery. Active gas aspiration provided a significantly superior effect on postoperative shoulder pain relief after diagnostic laparoscopy when compared to simple gas evacuation, without any adverse events. [9] In another study numerical pain intensity scale (NPIS) at the 24th h were significantly lower in Group 1 (p < 0.001). However, there were no significant differences in the NPIS scores following the 1st h and the 3rd day. No differences were found in the operation time (p > 0.05). According to the correlation analysis between the operation time and NPIS scores between the groups, in Group 1 the duration of surgery was significantly proportional to NPIS24. All patients were discharged from the hospital on the 4th postoperative day. [10] Rationale: Identifying the most eﬀective technique for gas removal may have significant implications for patient care and healthcare costs. Furthermore, given the widespread use of laparoscopic cholecystectomy, this study may have broader implications for other laparoscopic procedures that require abdominal insuﬄation. So the objective of this study is to determine if there is a signiﬁcant diﬀerence in postoperative pain scores between patients who receive active gas aspiration versus those who receive simple compression following laparoscopic cholecystectomy.

OBJECTIVE: The aim of this study is to compare outcome of active aspiration versus simple compression to remove residual gas from abdominal cavity in reducing pain after laparoscopic cholecystectomy.

OPERATIONAL DEFINITIONS Simple Compression: In this group, diagnostic laparoscopies commenced with a 5 mm intraumbilical vertical incision, followed by placement of the first bladeless umbilical port trocar (using 5 mm XCEL). Warm CO2 gas insufflation will create the pneumoperitoneum at a flow rate of 1-2.5 L/min; intra-abdominal pressure will be set at 12 mmHg. Patients will then placed in the Trendelenburg position (45°) and the second trocars (using 5 mm XCEL) will be placed at the suprapubic area. Chromopertubation with methylene blue will be performed, with electrocauterization of the endometriotic lesions if necessary. CO2 insufflation will be then ceased and all trocars will be opened. The surgeon will apply abdominal pressure to evacuate any residual CO2. The patient will be then placed in a neutral (horizon plane) position, the trocars will be removed and the incision closed.

Active Gas Aspiration: Once the trocars will be opened, aspiration cannula will be then placed through the accessory port reach at the subdiaphragmatic under direct visualization. After cessation of CO2 insufflation, residual gas will be removed by suctioning with 100 mmHg of pressure until the infra-diaphragmatic area of the abdominal wall close to liver surface. Negative pressure will be then ceased and the aspiration cannula will be taken out under direct vision. The procedure will be completed using the same method as the simple compression group.

Post-operative Pain: Patients' postoperative pain will be evaluated using a visual analogue scale (VAS) at the 1st, 4th and 12th postoperative hours by a surgical nurse. Pain severity will be assessed from 0 (no pain) to 10 (unbearable pain intensity). Daily analgesic requirements will be calculated in terms of consumption per day (Diclofenac sodium/bulb, 75 mg/ amp). Analgesics will be administered to patients whose VAS score will be more than 5.

HYPOTHESIS There is a difference in the outcome of active aspiration versus simple compression to remove residual gas from abdominal cavity in reducing pain after laparoscopic cholecystectomy.

MATERIALS AND METHODS Study Design: Comparative study Setting: East Surgical Ward, Mayo Hospital, Lahore. Duration of Study: Six months after approval of synopsis. Sample Size: 62 cases in each group were calculated by taking 5 % level of significance and 80% power of study with expected population proportion of analgesics requirement 43.2% in active gas aspiration group versus 67.6% in simple compression group (p value < 0.001). [9] Sampling Technique: Simple random sampling technique

SAMPLE SELECTION

Inclusion criteria:

* Patients of both genders.
* Patients of age ≥ 18 years.
* All patients presenting for elective laparoscopic cholecystectomy.

Exclusion Criteria:

* Patients suffering from obstructive jaundice anamnesis.
* Patients who had received a diagnosis of gallbladder cancer.
* Patients whose procedures were converted to open cholecystectomy during the surgery.
* Patients who had additional pathologies such as bronchial asthma, chronic obstructive pulmonary disease.
* Patients refused to give consent. DATA COLLECTION TOOLS After taking permission from hospital ethical committee 62 patients following inclusion criteria will be enrolled in this study. These patients will be divided into two groups by simple random sampling 31 in Group A (Active gas aspiration) and 31 in Group B (Simple compression). Informed consent will be taken from all the patients.

Quantitative and qualitative variables will be entered to the predesigned performa which is attached as appendix. Data on patient characteristics will be collected, including age, gender, height, weight, BMI, operation time, Used CO2, VAS score of shoulder pain at 1st, 4th, and 12th hour, and VAS score of abdominal pain at 1st, 4th, and 12th.

DATA ANALYSIS PROCEDURE:

Data will be entered to the SPSS version 20.00. Quantitative variables like age, height, weight, BMI, operation time, Used CO2, VAS score of shoulder pain at 1st, 4th, and 12th hour, and VAS score of abdominal pain at 1st, 4th, and 12th will be presented as mean ± standard deviation. Qualitative variables like gender and requirement of analgesics will be presented in form of frequency and percentage in both groups. Paired sample t-test will be applied to compare VAS score of shoulder pain at 1st, 4th, and 12th hour, and VAS score of abdominal pain at 1st, 4th, and 12th. Chi-square test will be applied to compare requirement of analgesics. P ≤ 0.05 will be considered as significant. Data will be stratified for age, gender and VAS score of shoulder pain at 1st, 4th, and 12th hour, and VAS score of abdominal pain at 1st, 4th, and 12th.

REFERENCES:

1. Mannam R, Narayanan RS, Bansal A, Yanamaladoddi VR, Sarvepalli SS, Vemula SL, Aramadaka S. Laparoscopic Cholecystectomy Versus Open Cholecystectomy in Acute Cholecystitis: A Literature Review. Cureus. 2023 Sep 21;15(9).
2. Khalid A, Khalil K, Qadri HM, Ahmad CZ, Fatima W, Raza A, Asif MA, Luqman MS, Nizami MF. Comparison of postoperative complications of open versus laparoscopic cholecystectomy according to the modified Clavien-Dindo Classification System. Cureus. 2023 Aug 17;15(8).
3. Park SJ. Postoperative shoulder pain after laparoscopic surgery. Journal of Minimally Invasive Surgery. 2020 Mar 3;23(1):3.
4. Özgönül A, Yalçın M, Öter V, Tatlı F, Yücel Y. The relationship between early postoperative pain and intraperitoneal residual gas after laparoscopic cholecystectomy. Laparoscopic Endoscopic Surgical Science (LESS).;25(2):59-63.
5. Riedel HH, Semm K. The post-laparoscopic pain syndrome (author's syndrome) [Article in German]. Geburtshilfe Frauenheilkd 1980;40:635-43.
6. Sao CH, Chan-Tiopianco M, Chung KC, Chen YJ, Horng HC, Lee WL, Wang PH. Pain after laparoscopic surgery: Focus on shoulder-tip pain after gynecological laparoscopic surgery. Journal of the Chinese Medical Association. 2019 Nov 1;82(11):819-26.
7. Umano GR, Delehaye G, Noviello C, Papparella A. The "dark side" of pneumoperitoneum and laparoscopy. Minimally Invasive Surgery. 2021 May 19;2021:1-9.
8. Rosenberg J, Fuchs-Buder T. Low-pressure pneumoperitoneum-why and how. Laparoscopic Surgery. 2023 Oct 30;7.
9. Leelasuwattanakul N, Bunyavehchevin S, Sriprachittichai P. Active gas aspiration versus simple gas evacuation to reduce shoulder pain after diagnostic laparoscopy: a randomized controlled trial. Journal of Obstetrics and Gynaecology Research. 2016 Feb;42(2):190-4.
10. Erdem H, Gençtürk M, Çetinkünar S, Şişik A, Sözen S. The effect of active gas aspiration to reduce pain after laparoscopic sleeve gastrectomy for morbid obesity: a randomized controlled study. Archives of Medical Science-Civilization Diseases. 2021;6(1):109-16.

ELIGIBILITY:
Inclusion criteria:

* Patients of both genders.
* Patients of age ≥ 18 years.
* All patients presenting for elective laparoscopic cholecystectomy.

Exclusion Criteria:

* Patients suffering from obstructive jaundice anamnesis.
* Patients who had received a diagnosis of gallbladder cancer.
* Patients whose procedures were converted to open cholecystectomy during the surgery.
* Patients who had additional pathologies such as bronchial asthma, chronic obstructive pulmonary disease.
* Patients refused to give consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2025-12-11 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2027-01-30 (Estimated)

PRIMARY OUTCOMES:
Numerical Pain Intensity Scale (NPIS) | 24 hours
  The Numerical Pain Intensity Scale (NPIS) is a simple, self-reported tool commonly used in clinical settings to assess the intensity of a person's pain. It typically ranges from 0 to 10, with 0 indicating "no pain" and 10 representing "the worst pain imaginable." Patients are asked to rate their pain based on their current experience, providing healthcare professionals with a clear indication of the pain's severity. This scale is useful for tracking pain changes over time, evaluating the effectiveness of treatments, and facilitating communication between patients and providers about pain management. The NPIS is valued for its ease of use and ability to provide quick, quantifiable insights into a patient's pain level.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Erdem H, Gençtürk M, Çetinkünar S, Şişik A, Sözen S. The effect of active gas aspiration to reduce pain after laparoscopic sleeve gastrectomy for morbid obesity: a randomized controlled study. Archives of Medical Science-Civilization Diseases. 2021;6(1):109-16.
- [Result] Leelasuwattanakul N, Bunyavehchevin S, Sriprachittichai P. Active gas aspiration versus simple gas evacuation to reduce shoulder pain after diagnostic laparoscopy: A randomized controlled trial. J Obstet Gynaecol Res. 2016 Feb;42(2):190-4. doi: 10.1111/jog.12868. Epub 2015 Dec 3. PMID 26633582
- [Result] Rosenberg J, Fuchs-Buder T. Low-pressure pneumoperitoneum-why and how. Laparoscopic Surgery. 2023 Oct 30;7.
- [Result] Umano GR, Delehaye G, Noviello C, Papparella A. The "Dark Side" of Pneumoperitoneum and Laparoscopy. Minim Invasive Surg. 2021 May 19;2021:5564745. doi: 10.1155/2021/5564745. eCollection 2021. PMID 34094598
- [Result] Sao CH, Chan-Tiopianco M, Chung KC, Chen YJ, Horng HC, Lee WL, Wang PH. Pain after laparoscopic surgery: Focus on shoulder-tip pain after gynecological laparoscopic surgery. J Chin Med Assoc. 2019 Nov;82(11):819-826. doi: 10.1097/JCMA.0000000000000190. PMID 31517775
- [Result] Özgönül A, Yalçın M, Öter V, Tatlı F, Yücel Y. The relationship between early postoperative pain and intraperitoneal residual gas after laparoscopic cholecystectomy. Laparoscopic Endoscopic Surgical Science (LESS).;25(2):59-63.
- [Result] Park SJ. Postoperative Shoulder Pain after Laparoscopic Surgery. J Minim Invasive Surg. 2020 Mar 15;23(1):3-4. doi: 10.7602/jmis.2020.23.1.3. PMID 35600729
- [Result] Khalid A, Khalil K, Mehmood Qadri H, Ahmad CZ, Fatima W, Raza A, Asif MA, Luqman MS, Jawariah, Nizami MFK. Comparison of Postoperative Complications of Open Versus Laparoscopic Cholecystectomy According to the Modified Clavien-Dindo Classification System. Cureus. 2023 Aug 17;15(8):e43642. doi: 10.7759/cureus.43642. eCollection 2023 Aug. PMID 37727181
- [Result] Mannam R, Sankara Narayanan R, Bansal A, Yanamaladoddi VR, Sarvepalli SS, Vemula SL, Aramadaka S. Laparoscopic Cholecystectomy Versus Open Cholecystectomy in Acute Cholecystitis: A Literature Review. Cureus. 2023 Sep 21;15(9):e45704. doi: 10.7759/cureus.45704. eCollection 2023 Sep. PMID 37868486